CLINICAL TRIAL: NCT01754142
Title: Kombiglyze XR (Saxagliptin + Metformin XR Fixed Dose Combination) Regulatory Postmarketing Surveillance
Brief Title: Korean Post-marketing Surveillance for Kombiglyze XR®
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: CV181-306
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 2 diabetes mellitus subjects initiating Kombiglyze XR: Patients with diagnosis of type 2 diabetes mellitus initiating Kombiglyze XR treatment within the approved indications will be enrolled

SUMMARY:
The purpose of this post-marketing surveillance is to investigate and confirm the type and incidence of newly identified adverse events and any other factors affecting safety and efficacy of Kombiglyze Extended release (XR) so that the regulatory authority can manage the marketing approval properly

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* ≥ 18 years of age
* Have diagnosed Type 2 diabetes mellitus (T2DM)
* Are initiating Kombiglyze XR treatment within the approved Korean indications

Exclusion Criteria:

* Being treated for an indication not approved for the use of Kombiglyze XR in Korea
* Is contraindicated for the use of Kombiglyze XR as described in the Korean label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of type 2 diabetes mellitus initiating Kombiglyze XR treatment within the approved indications will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 755 (Actual)
Dates: Start 2012-11-24 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of known and unexpected adverse events, especially serious adverse events | 30 days after last dose of study drug (Approximately up to 4.5 years)
Incidence of adverse events under the routine drug use | 30 days after last dose of study drug (Approximately up to 4.5 years)
Effectiveness of Kombiglyze XR as assessed by change from baseline in Hemoglobin A1c (HbA1c), Fasting plasma glucose (FPG), and 2-hour post-prandial glucose (2-hr PPG) | Baseline and Week 12
Effectiveness of Kombiglyze XR as assessed by change from baseline in Hemoglobin A1c (HbA1c), Fasting plasma glucose (FPG), and 2-hour post-prandial glucose (2-hr PPG) | Baseline and Week 24 (for patients that have a post Week 12 follow-up visit)

SECONDARY OUTCOMES:
Safety information related to factors (eg, gender, demographics etc) that may affect the safety of the drug based on incidence rates of AEs | Approximately up to 4.5 years
  Adverse events (AEs)
Safety information related to factors (eg, gender, demographics etc) that may affect the effectiveness of the drug based on incidence rates of AEs | Approximately up to 4.5 years
Safety information related to overdose, drug-to-drug interaction and laboratory abnormalities based on incidence rates of AEs | Approximately up to 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Research Site, Seoul, South Korea

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4126&filename=CSR_Synopsis_CV181_306.pdf